CLINICAL TRIAL: NCT07374120
Title: Treatment Patterns and Key Endpoints Among Patients With Chronic-Phase Chronic Myeloid Leukemia (CML-CP) in a Community Oncology Setting
Brief Title: Treatment Patterns and Key Endpoints Among Patients With Chronic-Phase Chronic Myeloid Leukemia in a Community Oncology Setting
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A0US12
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
Keywords: CML; Tyrosine kinase inhibitors; Treatment patterns; Real-world
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- CML-CP Group: Patients with a diagnosis of CML-CP who initiated 1L TKI treatment in The US Oncology Network practices between 01 January 2016 and 31 December 2022.

SUMMARY:
This was a retrospective observational study to examine treatment patterns, molecular testing patterns, treatment response, and clinical outcomes among patients initiating first-line (1L) tyrosine kinase inhibitor (TKI) treatment for CML-CP in The United States (US) Oncology Network practices.

Patients who initiated 1L therapy between 01 January 2016 and 31 December 2022 were eligible for inclusion in the study. Study-eligible patients were followed longitudinally post-index until death (if the patient had documentation of death during the study observation period) or last available patient record that occurred on or before the end of the study observation period. The study observation period was from 01 January 2016 to 30 November 2023. The index date was defined as the start date of 1L therapy for CML-CP.

ELIGIBILITY:
Inclusion criteria:

1. Patients whose data were accessible for research purposes during the study observation period.
2. Patients diagnosed with CML-CP at first recorded diagnosis of CML.
3. Patients ≥ 18 years of age at first recorded diagnosis of CML.
4. Patients who initiated qualifying 1L therapy for CML-CP during the study identification period. Qualifying 1L therapy treatments consisted of imatinib, dasatinib, bosutinib, or nilotinib as monotherapy.
5. Patients with ≥1 visit within The US Oncology Network practices following initiation of 1L therapy and through the end of the study observation period.

Exclusion criteria:

1. Patients enrolled in interventional clinical trials during the study observation period.
2. Patients who received any systemic treatment indicated for another primary cancer during the study observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1480 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Time From Initial CML Diagnosis to Initiation of 1L TKI Treatment | Baseline
Number of Patients who Received a Stem Cell Transplant (SCT) | Up to approximately 7 years
Number of Patients by Type of 1L and Second-line (2L) TKI Treatment | Up to approximately 7 years
Number of Patients by Initial Dose of Each TKI in 1L and 2L Treatment | Up to approximately 7 years
Number of Patients by Treatment Sequence From 1L TKI to 2L TKI Treatment | Up to approximately 7 years
Number of Patients by Dose Modification of 1L and 2L TKI Treatment | Up to approximately 7 years
  Dose modifications included dose escalation, reduction, or hold.
Number of Patients by Reason for Dose Modification of 1L and 2L TKI Treatment | Up to approximately 7 years
  Dose modifications included dose escalation, reduction, or hold.
Number of Patients who Discontinued 1L and 2L TKI Treatment | Up to approximately 7 years
Number of Patients by Reason for Discontinuing 1L and 2L TKI Treatment | Up to approximately 7 years
Number of Patients by Clinical Events of Interest During 1L and 2L TKI Treatment | Up to approximately 7 years
  Clinical events of interest included:
  * Alopecia
  * Anemia
  * Arthralgia/Myalgia
  * Diarrhea
  * Elevated liver enzyme
  * Elevated serum creatinine
  * Fatigue
  * Febrile neutropenia
  * Infection secondary to neutropenia
  * Interstitial lung disease-like events
  * Leukopenia
  * Nausea
  * Neutropenia
  * Pain
  * Prolongation of QT interval
  * Thrombocytopenia
  * Venous embolism (including pulmonary embolism and/or deep vein thrombosis)
  * Vomiting
Number of Patients by Best Overall Molecular Response (MR) Achieved During 1L and 2L TKI Treatment | Up to approximately 7 years
  MR was based on BCR::ABL (International Scale [IS]) qPCR testing results. Molecular response was categorized as:
  * MR 2: if BCR::ABL (IS) >0.1% - ≤ 1%
  * Major MR (MMR)/MR 3: if BCR::ABL(IS) >0.01% - ≤0.1%
  * MR 4: if BCR::ABL1 (IS) >0.0032% -≤0.01%
  * MR 4.5: if BCR::ABL (IS) ≤0.0032%
  * Not documented
Number of Patients by Best Overall MR Achieved Within 12 Months of Initiating 1L and 2L TKI Treatment | From Baseline up to 12 months
  MR was based on BCR::ABL (IS) qPCR testing results. Molecular response was categorized as:
  * MR 2: if BCR::ABL (IS) >0.1% - ≤ 1%
  * Major MR (MMR)/MR 3: if BCR::ABL(IS) >0.01% - ≤0.1%
  * MR 4: if BCR::ABL1 (IS) >0.0032% -≤0.01%
  * MR 4.5: if BCR::ABL (IS) ≤0.0032%
  * Not documented
Number of Patients by MR Achieved After Initiating 1L and 2L TKI Treatment | 6, 12, 18, and 24 months
  MR was based on BCR::ABL (IS) qPCR testing results. Molecular response was categorized as:
  * MR 2: if BCR::ABL (IS) >0.1% - ≤ 1%
  * Major MR (MMR)/MR 3: if BCR::ABL(IS) >0.01% - ≤0.1%
  * MR 4: if BCR::ABL1 (IS) >0.0032% -≤0.01%
  * MR 4.5: if BCR::ABL (IS) ≤0.0032%
  * Not documented
Number of Patients who Achieved a BCR::ABL (IS) Result ≤10% Within 6 Months of Initiating 1L and 2L TKI Treatment | From Baseline up to 6 months
Number of Patients who Achieved or Sustained a BCR::ABL (IS) Result <1% Between 6 and 12 Months After Initiating 1L and 2L TKI Treatment | From Month 6 to Month 12
Number of Patients who Achieved or Sustained a BCR::ABL (IS) Result ≤0.1% Between 13 and 24 Months After Initiating 1L and 2L TKI Treatment | From Month 13 to Month 24
Number of Patients who Achieved or Sustained a BCR::ABL (IS) Result ≤0.1% After 24 Months Following Initiating 1L and 2L TKI Treatment | From Month 24 to end of study, up to approximately 6 years
Number of Patients who Achieved Complete Hematologic Response (CHR) During 1L and 2L TKI Treatment | Up to approximately 7 years
  CHR was observed when white blood cells, hemoglobin, and platelet counts were all within each respective normal lab range.
Number of Patients who Achieved CHR Within 12 Months of Initiating 1L and 2L TKI Treatment | From Baseline up to 12 months
  CHR was observed when white blood cells, hemoglobin, and platelet counts were all within each respective normal lab range.
Number of Patients who Achieved Complete Cytogenetic Response (CCyR) During 1L and 2L TKI Treatment | Up to approximately 7 years
  Cytogenetic response was based on the Philadelphia chromosome results. CCyR was defined as having no Philadelphia chromosome-positive metaphases.
Number of Patients who Achieved CCyR Within 12 Months of Initiating 1L and 2L TKI Treatment | From Baseline up to 12 months
  Cytogenetic response was based on the Philadelphia chromosome results. CCyR was defined as having no Philadelphia chromosome-positive metaphases.
Duration of Therapy (DOT) for 1L TKI Treatment | Up to approximately 7 years
  DOT was defined as the interval between the start date of the 1L therapy (index date) and the end date of 1L therapy, including any treatment interruptions or other breaks.
DOT for 2L TKI Treatment | Up to approximately 7 years
  DOT was defined as the interval between the start date of the 2L therapy and the end date of 2L therapy, including any treatment interruptions or other breaks.
Progression-free Survival (PFS) for 1L TKI Treatment | Up to approximately 7 years
  PFS was defined as physician-documented progression, loss of MR2, BCR::ABL (IS) ≤1%, or an increase in BCR::ABL1 transcript to >1%, or a 1-log increase in BCR::ABL1 transcript levels with loss of MMR.
PFS for 2L TKI Treatment | Up to approximately 7 years
  PFS was defined as physician-documented progression, loss of MR2, BCR::ABL (IS) ≤1%, or an increase in BCR::ABL1 transcript to >1%, or a 1-log increase in BCR::ABL1 transcript levels with loss of MMR.
Overall Survival (OS) for 1L TKI Treatment | Up to approximately 7 years
  OS was defined as the interval between the start date of 1L therapy (index date) and the date of death (any cause).
Overall Survival (OS) for 2L TKI Treatment | Up to approximately 7 years
  OS was defined as the interval between the start date of 2L therapy and the date of death (any cause).
Treatment-free Interval (TFI) | Up to approximately 7 years
  TFI was defined as the interval between the discontinuation date of 1L therapy and the start date of 2L therapy or date of death.

SECONDARY OUTCOMES:
Number of Patients With BCR::ABL Testing (per National Comprehensive Cancer Network (NCCN) Guidelines) at Diagnosis | Baseline
Number of Patients With BCR::ABL Testing (per NCCN Guidelines) in 3-Month Intervals After Initiation of 1L and 2L TKI Treatment Until BCR::ABL1 ≤1% was Achieved | Up to approximately 7 years
After Initiation of 1L and 2L TKI Treatment, Number of Patients With BCR::ABL Testing (per NCCN Guidelines) in 3-Month Intervals Within 2 Years After BCR::ABL1 ≤1% was Achieved | 2 years
After Initiation of 1L and 2L TKI Treatment, Number of Patients With BCR::ABL Testing (per NCCN Guidelines) Between 1 and 3 Months Following 2 Years After BCR::ABL1 ≤1% was Achieved | Up to approximately 5 years
Number of BCR::ABL Tests (per NCCN Guidelines) After Initiation of 1L and 2L TKI Treatment Until BCR::ABL1 ≤1% was Achieved | Up to approximately 7 years
Following Initiation of 1L and 2L TKI Treatment, Number of BCR::ABL Tests (per NCCN Guidelines) Within 2 Years After Achieving BCR::ABL1 ≤1% | 2 years
Following Initiation of 1L and 2L TKI Treatment, Number of BCR::ABL Tests (per NCCN Guidelines) Performed After 2 Years of Achieving BCR::ABL1 ≤1% | Up to approximately 5 years
Number of Patients With BCR::ABL Testing (per European LeukemiaNet (ELN) Guidelines) at Diagnosis | Baseline
Number of Patients With BCR::ABL Testing (per ELN Guidelines) in 3-Month Intervals After Initiation of 1L and 2L TKI Treatment Until BCR::ABL1 ≤0.1% was Achieved | Up to approximately 7 years
Number of Patients With BCR::ABL Testing (per ELN Guidelines) Tested in 3-Month Intervals After Initiation of 1L Until BCR::ABL1 ≤0.1% was Achieved and Tested Between 2 to 6 Months Until CCyR was Achieved | 5 months
Number of Patients With BCR::ABL Testing (per ELN Guidelines) Tested in 3-Month Intervals After Initiation of 2L Until BCR::ABL1 ≤0.1% was Achieved and Tested Between 2 to 6 Months Until CCyR was Achieved | 5 months
Number of Patients With BCR::ABL Testing (per ELN Guidelines) Tested in 3-Month Intervals After Initiation of 1L Until BCR::ABL1 ≤0.1% was Achieved and Tested Every 12 Months Until CCyR was Achieved | Up to approximately 7 years
Number of Patients With BCR::ABL Testing (per ELN Guidelines) Tested in 3-Month Intervals After Initiation of 2L Until BCR::ABL1 ≤0.1% was Achieved and Tested Every 12 Months Until CCyR was Achieved | Up to approximately 7 years
Number of BCR::ABL Tests (per ELN Guidelines) After Initiation of 1L and 2L TKI Treatment Until BCR::ABL1 ≤0.1% was Achieved | Up to approximately 7 years
Number of BCR::ABL Tests (per ELN Guidelines) After Initiation of 1L and 2L TKI Treatment Until CCyR was Achieved | Up to approximately 7 years
Number of Molecular Testing by Year Following Initiation of 1L TKI Treatment During Which the T315I Mutation was Identified | Up to approximately 7 years
Number of Patients With T3151 Mutation Testing During 1L and 2L TKI Treatment | Up to approximately 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18406